CLINICAL TRIAL: NCT00976326
Title: A Trial Investigating the Pharmacokinetic and Safety Profiles of NN1250 in Subjects With Mild, Moderate and Severe Degrees of Hepatic Impairment and in Subjects With Normal Hepatic Function
Brief Title: A Trial Investigating the Pharmacokinetic (Mode of Action in the Body) and Safety Profiles of NN1250 (Insulin Degludec) in Subjects With Various Degrees of Impaired Liver Function and in Subjects With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-1989; 2009-009465-34 (EudraCT Number)
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: Healthy volunteers (Experimental)
  Interventions: Drug: insulin degludec
- B: Subjects with mild liver impairment (Experimental)
  Interventions: Drug: insulin degludec
- C: Subjects with moderate liver impairment (Experimental)
  Interventions: Drug: insulin degludec
- D: Subjects with severe liver impairment (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — The dose level will be one single dose of 0.4 units per kg body weight injected s.c. (subcutaneously, under the skin)

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to evaluate if the pharmacokinetic and safety profiles of NN1250 (insulin degludec) are altered to such an extent that the dose should be adjusted in subjects with impaired liver function compared to the dose for subjects with normal liver function.

ELIGIBILITY:
Inclusion Criteria:

* Subject with normal hepatic function, liver parameters within normal range. Not assessed with the Child-Pugh criteria. Or: Subject with stable hepatic impairment classified as Child-Pugh grade A, B or C as assessed by Investigator
* Body mass index maximum 40.0 kg/m^2

Exclusion Criteria:

* Subject with any disease or condition which the Investigator feels would interfere with the trial outcome or execution except for conditions associated with hepatic impairment in the group of subjects with compromised hepatic function
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Not able or willing to refrain from smoking during the inpatient period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Area under the NN1250 concentration-time curve after single-dose | from 0 to 120 hours

SECONDARY OUTCOMES:
Maximum observed NN1250 concentration after single-dose | from 0 to 120 hours
Renal clearance of NN1250 | from 0 to 24 hours
Number of adverse events | from Visit 2, Day -1 until Follow-up Visit

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Result] Kupcova V, Arold G, Roepstorff C, Hojbjerre M, Klim S, Haahr H. Insulin degludec: pharmacokinetic properties in subjects with hepatic impairment. Clin Drug Investig. 2014 Feb;34(2):127-33. doi: 10.1007/s40261-013-0154-1. PMID 24277680
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com